CLINICAL TRIAL: NCT01884493
Title: Electrophysiological Investigation and rTMS Intervention of Ambulatory Central Processing of Freezing of Gait in Parkinson's Disease
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Principal Investigator, Chon-Haw Tsai, The chief, Department of Neurology, China Medical University Hospital
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: CMUH102-REC1-002
Record Dates: First submitted 2013-06-19; First posted 2013-06-24 (Estimated); Last update posted 2014-08-08 (Estimated); Status verified 2014-01

CONDITIONS: Parkinson's Disease; Parkinson's Disease With Freezing of Gait
Keywords: Parkinson's Disease; Freezing of Gait; movement-related cortical potential; repetitive transcranial magnetic stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- real iTBS (Experimental): The paradigm will use a theta burst stimulation pattern (TBS) in which 3 pulses of stimulation will be given at 50Hz, repeated every 200 ms. In the iTBS, a 2-second train of TBS is repeated every 10 seconds for a total of 190 seconds (600 pulses). Subjects will be 8 courses of iTBS stimulation in 10 business days.
  Interventions: Device: real iTBS; Device: sham iTBS
- sham iTBS (Sham Comparator): Subjects will be 8 courses of sham iTBS stimulation in 10 business days.
  Interventions: Device: real iTBS; Device: sham iTBS

INTERVENTIONS:
Device: real iTBS — Theta-burst magnetic stimulation (TBS) is a repetitive transcranial magnetic stimulation (rTMS) technique that elicits long-lasting changes in the excitability of human primary motor cortex (M1).
Device: sham iTBS — The sham test will be done by transferring the double cone coil 90 degrees anteriorly and putting the lower edge of the coil of the vertex.

SUMMARY:
The gait symptoms are usually refractory to the dopaminergic agents and some other resolutions, i.e. repetitive transcranial magnetic stimulation (rTMS) should be searched for in this regard. To study the impact of rTMS, investigators will adopt a domestically developed ambulatory recorder (PK-16CH EXG) for the concomitant recording of the electroencephalographic and electromyographic signals for PD patients when walking in the gait laboratory or when conducting leg dorsiflexion movement on sitting.

DETAILED DESCRIPTION:
The Bereitschaftspotential (BP), event related synchronization (ERS) and event related dysynchronization (ERD) will be analyzed for the investigation of the possible differences of brain activities prior to leg voluntary movement between patients and controls. In addition, the synchronized recorded gait parameters for gait ignition,turning and termination will also be analyzed. The information gathered will allow us to further understand the pathophysiology of the gait freezing in PD. Investigators will deliver a course of rTMS with intermittent theta burst paradigm of the leg motor cortex to investigate whether the non-invasive brain stimulation can ameliorate the gait freezing in PD patients. The subjects will be assessed before and 4 times after rTMS during an 8-week period with clinical scoring batteries and electrophysiological recording as aforementioned. At the end of the 8th week, the test group and sham group will cross over and undergo the same procedures as aforementioned. The serial comprehensive investigations in this project will not only promote our understanding of the gait freezing pathophysiology but also may charge a novel trail for the management of long suffering symptom of the PD patients.

ELIGIBILITY:
Inclusion Criteria:

Patients with PD will be diagnosed according to the Brain Bank criteria.

Exclusion Criteria:

1. Patients had past history of epilepsy, intracranial operation or brain tumor.
2. Hoehn & Yahr Stage V.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Change in Laboratory gait analysis after 8 courses of iTBS | baseline to week 8
  Variables in gait analysis:1.Gait initiation; 2.Level walking; 3.Turning; 4.Gait termination.

SECONDARY OUTCOMES:
Change in Unified Parkinson's Disease Rating Scale (UPDRS) after 8 courses of iTBS | baseline to week 8
Change in The 39-item Parkinson's Disease Questionnaire (PDQ-39) after 8 courses of iTBS | baseline to week 8
Change in Fall assessment test after 8 courses | baseline to week 8
Change in Tinetti's Mobility Index after 8 courses of iTBS | baseline to week 8
Change in new freezing of gait questionnaire (FOG-Q) after 8 courses | baseline to week 8
Change in Patients' Global Impressions of Change (PGIC) Scale after 8 courses of iTBS | baseline to week 8
Change in Clinical Global Impressions (CGI) after 8 courses of iTBS | baseline to week 8

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital/Neuro Depart, Taichung, Taiwan